CLINICAL TRIAL: NCT03598426
Title: Conventional Prophylactic Regimen of Oral Dexamethasone Versus Short-course Intravenous Dexamethasone in Preventing Paclitaxel-related Hypersensitivity Reactions in Breast and Gynecologic Oncology Patients
Brief Title: Conventional Prophylactic Oral Dexamethasone vs Short-course IV Dexamethasone in Paclitaxel Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Linda Hong, MD, Primary Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5180198
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Hypersensitivity Reactions
MeSH Terms: conditions — Hypersensitivity | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Single center, prospective, randomized, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional (Active Comparator): Oral dexamethasone (20 mg) at home, 12 hours and 6 hours prior to paclitaxel infusion. On the day of treatment at the clinic, an intravenous administration of diphenhydramine 50 mg and famotidine 20 mg, administered 30 minutes prior to paclitaxel infusion.
  Interventions: Drug: Dexamethasone
- Short-Course (Active Comparator): Intravenous administration of dexamethasone 20 mg, along with an intravenous administration of diphenhydramine 50 mg and famotidine 20 mg, administered 30 minutes prior to paclitaxel infusion.
  Interventions: Drug: Dexamethasone
- Combined (Active Comparator): Oral dexamethasone (20 mg) at home, 12 hours prior to paclitaxel infusion. On the day of treatment at the clinic, an additional intravenous administration of dexamethasone 20 mg, along with an intravenous administration of diphenhydramine 50 mg and famotidine 20 mg, administered 30 minutes prior to paclitaxel infusion.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Conventional arm will only use oral dexamethasone as intervention; Short-Course arm will only use intravenous dexamethasone as intervention; Combined arm will use both oral and intravenous dexamethasone as intervention
  Other Names: Decadron

SUMMARY:
This study is a single center, prospective, randomized, open-label study aimed at determining the most effective means of preventing hypersensitivity reactions in gynecologic oncology patients receiving paclitaxel infusions. The study will therefore provide clinicians with the best ways of preventing paclitaxel hypersensitivity reactions in their patients during treatment. Subjects will be randomized using the block randomization method into one of these three commonly used treatment methods:(1) Conventional method: oral dexamethasone (20 mg), taking 12 hours and 6 hours prior to paclitaxel infusion and intravenous administration of histamine-1 (H1), and a histamine-2 (H2)receptor antagonists administered 30 minutes prior to paclitaxel infusion. (2) Short-course method: intravenous dexamethasone (20 mg), administered concurrently with H1 and H2 antagonists, 30 minutes prior to paclitaxel infusion. (3) Combined method: oral dexamethasone (20 mg), taking 12 hours prior to treatment in addition to intravenous dexamethasone (20 mg), H1 and H2 receptor antagonists administered 30 minutes prior to paclitaxel infusion. The one-way analysis of variance (ANOVA) would be used to determine if there is any significant difference between the different strategies that are used to pre-medicate patients prior to paclitaxel infusion. P-values of less than 0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
One of the potentially serious and dose-limiting toxicities of paclitaxel is the development of hypersensitivity reactions (HSRs). Up to 42% of patients receiving paclitaxel experience an HSR, with serious (> grade 3) reactions observed in about 2% of patients. Paclitaxel prescribing information and many other references therefore strongly recommend pre-medicating patients who are to be treated with paclitaxel-containing regimen with a corticosteroid, a histamine-1 (H1), and a histamine-2 (H2) antagonist prior to paclitaxel infusion. This is done to help prevent or minimize the occurrence of HSRs that could be caused by treating patients with paclitaxel. However, the method and timing of administering these pre-medications (particularly in the case of dexamethasone) have not been standardized. The current and most commonly used methods of preventing paclitaxel HSR includes one of the following: 1. Administering oral dexamethasone (20 mg), 12 hours and 6 hours prior to paclitaxel infusion and intravenous administration of H1 and H2 receptor antagonists 30 minutes prior to paclitaxel infusion (Conventional method); 2. Administering intravenous dexamethasone (20 mg), concurrently with H1 and H2 antagonists, 30 minutes prior to paclitaxel infusion (Short-course method); 3. Administering oral dexamethasone (20 mg), 12 hours prior to treatment in addition to intravenous dexamethasone (20 mg), H1 and H2 receptor antagonists administered 30 minutes prior to paclitaxel infusion. The goal of this study is to do a single center, prospective, randomized, open-label study to determine the most effective method in preventing paclitaxel HSR among these three commonly used methods.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients > 18 years of age
2. Patients of the Loma Linda University Health (LLUH) gynecologic oncology and breast oncology service
3. Confirmed breast or gynecologic cancer diagnosis of any stage and any gynecologic or breast malignancy
4. Planned treatment with paclitaxel containing regimen either in the adjuvant setting or for palliation
5. Planned treatment with paclitaxel should be for 3 or more cycles given as a weekly or every 3 weeks cycle
6. Paclitaxel should be given as a monotherapy or as part of a combination regimen. If paclitaxel is part of a regimen containing other drugs, the following conditions must be met:

   1. Paclitaxel will be the first chemotherapy regimen to be infused when patient comes in for treatment
   2. Chemotherapy regimen that would be approved for the study are the following:

   i. Paclitaxel/ Carboplatin ii. Paclitaxel/Carboplatin/Bevacizumab iii. Paclitaxel/Cisplatin/Bevacizumab iv. Paclitaxel/Bevacizumab v. Paclitaxel/ Ifosfamide vi. Paclitaxel/ Pazopanib
7. Patients should have no prior exposure to taxanes (this includes: paclitaxel, docetaxel, and protein-bound paclitaxel)
8. The chemotherapy treatment should be at one of the LLUH Adult Cancer Centers
9. The patient should be an English or Spanish speaking patient

Exclusion Criteria:

1. Patients who are not with the gynecologic or breast oncology service
2. Patients who are with the gynecologic oncology or breast oncology service but are not receiving paclitaxel either as a monotherapy or in combination with other regimen
3. Patients who have had prior exposure to taxanes (this includes: paclitaxel, docetaxel, and protein-bound paclitaxel)
4. Patients who are currently on steroid therapy and it is anticipated that therapy will not be discontinued at least a week prior to start of chemotherapy
5. Patients with autoimmune diseases, malignancies, and any other co-morbid condition that might require steroid therapy during chemotherapy. This includes, but not limited to:

   1. Crohn's disease
   2. Immune thrombocytopenia
   3. Lupus nephritis
   4. Multiple sclerosis
   5. Primary brain tumors
   6. Multiple Myeloma
   7. Hodgkin's Lymphoma
6. Patients with uncontrolled diabetes or diabetic or pre-diabetic patients with baseline A1C levels > 8.5
7. Patients who are allergic to diphenhydramine and/or dexamethasone
8. Non-English and Non-Spanish speaking patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 90 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Least incidence of any-grade-paclitaxel-HSR first cycle | 1 to 3 HOURS
  The treatment group that had the least incidence of any-grade-paclitaxel-HSR in the first cycle of chemotherapy treatment

SECONDARY OUTCOMES:
Least incidence of any-grade-paclitaxel-HSR in the first and second cycles | 1 to 3 HOURS
  The treatment group that had the least incidence of any-grade-paclitaxel-HSR in the first and second cycles of chemotherapy treatment
Least incidence of grade 3 or more paclitaxel-HSR in the first and second cycles | 1 to 3 HOURS
  The treatment group that had the least incidence of grade 3 or more paclitaxel-HSR in the first and second cycles of chemotherapy treatment
Least incidence of any-grade-paclitaxel-HSR second cycle | 1 to 3 HOURS
  The treatment group that had the least incidence of any-grade-paclitaxel-HSR in the second cycle of chemotherapy treatment
Least incidence of grade 3 or more paclitaxel-HSR first cycle | 1 to 3 HOURS
  The treatment group that had the least incidence of grade 3 or more paclitaxel-HSR in the first cycle of chemotherapy treatment
Least incidence of grade 3 or more paclitaxel-HSR second cycle | 1 to 3 HOURS
  The treatment group that had the least incidence of grade 3 or more paclitaxel-HSR in the second cycle of chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hong, MD, Principal Investigator — Loma Linda University Cancer Center
Locations (1):
- Loma Linda University Cancer Center, Loma Linda, California, United States